CLINICAL TRIAL: NCT05722730
Title: Effects of Pilates in Patients With Post- -COVID-19 Syndrome: Controlled and Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michele de Aguiar Zacaria (Other)
Responsible Party: Sponsor-Investigator, Michele de Aguiar Zacaria, Principal Investigator, Centro Universitário Augusto Motta
Organization: Centro Universitário Augusto Motta (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTC12345678
Record Dates: First submitted 2022-10-24; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; Pilates Method; Functional Status; Health-related quality of life; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial involving participants, who have developed the severe form of COVID-19 and required at least 7 days of invasive mechanical ventilation. They will be previously randomized in a 1:1 ratio by electronic system and blindly allocated to the intervention group that will perform an exercise protocol based on the Pilates method, 2x/week, for 12 weeks in therapeutic sessions of identical protocols lasting 60 min. All patients will be evaluated before and after for six minutes walk distance test, peripheral and respiratory muscle strength and endurance, post-COVID-19 functional status, dyspnea, fatigue and quality of life. The analysis of the data obtained during the research was carried out by an independent statistician who had access to the coded data and were based on intention-to-treat principles.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Initial assessments and assessments relating to clinical evolution will be conducted by an assessor blinded to treatment allocation. The evaluator will undergo an in-depth evaluation training program. An employee outside the research team will feed the computer database into secretly coded spreadsheets so that the independent statistician and researchers can analyze the data without having access to allocation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): The Pilates exercise protocol was designed based on protocols contained in previously published clinical trials whose objective had been muscle strengthening or improvement of muscle fatigue. Thus, the protocol will perform exercises from the classic repertoire of the Pilates Method, using equipment exclusive to the Method - such as Cadillac, Lader Barrel, Chair and Reformer. The sessions will take place twice a week, in a group of up to 3 participants, always in the morning lasting 60 minutes, with 10 minutes of warm-up, 40 minutes of load exercises and 10 minutes of relaxation exercises and calm down. All sessions were carried out by a physiotherapist specialized in the method, in a specific outpatient clinic. The professional who conducted the Pilates sessions, performed the proposed protocol, is unaware of the outcomes studied by the project.
  Interventions: Procedure: Pilates Exercises
- Control (No Intervention): Only follow-up of the clinical evolution will be carried out

INTERVENTIONS:
Procedure: Pilates Exercises — The intervention group will perform an exercise protocol based on the Pilates method, by a physiotherapist specialized in Pilates and independent of the researchers, using the method's own equipment, with a frequency of 2x/week, for 12 weeks in therapeutic sessions of identical protocols lasting 60 min.
  Other Names: Therapeutic Pilates
  Arms: Pilates

SUMMARY:
The COVID-19 is closely related to severe acute respiratory syndrome (SARS) with direct and indirect effects on several systems, especially the musculoskeletal system, in addition to the respiratory system. Some of these symptoms persist for a long time, called Post-COVID-19 Syndrome, directly interfering with the functional capacity and quality of life of these patients. Pilates exercises focus on breathing, postural symmetry, trunk stabilization, flexibility, joint mobility and strengthening through the full range of motion of all joints and not isolated muscle groups. The objective of this study will be to evaluate the clinical and functional effects of a Pilates for patients post hospitalization for COVID-19. A randomized and controlled clinical trial will be conducted, with recruitment patients who have developed the severe form of COVID-19 and required at least 7 days of invasive mechanical ventilation. They will be previously randomized in a 1:1 ratio by electronic system and blindly allocated to the intervention group that will perform an exercise protocol based on the Pilates method, 2x/week, for 12 weeks in therapeutic sessions of identical protocols lasting 60 min. All patients will be evaluated before and after for six minutes walk distance test, peripheral and respiratory muscle strength and endurance, post-COVID-19 functional status, dyspnea, and quality of life. The analysis will be based on intention-to-treat principles. Descriptive statistics will be used to present the characteristics of participants in the two treatment groups. P values less than 0.05 will be considered to indicate statistical evidence of significance. The variables of dyspnea, peripheral and respiratory muscle strength, functional capacity, post-COVID functional status and HRQoL will be analyzed using linear models of repeated measures which included all values measured after randomization with baseline scores and treatment clusters as covariates. Adjusted mean differences will be tested 12 weeks after randomization and start of intervention. Multiple comparisons will be performed using the Tukey Test with p-values adjusted using the Holm procedure. Baseline variables will be evaluated as predictors and moderators of treatment effects, including terms and interaction models. Effect sizes for primary and secondary endpoints will be calculated as Cohen's d from estimated marginal means (SMD) and standard error estimates from the adjusted primary analysis. All analyzes were performed using RStudio version 0.99.486. Results: The expected results are based on the alternative hypothesis that Pilates exercises are clinically effective, improving functional performance, exercise tolerance, reducing symptoms and improving the quality of life of patients with symptoms of Post-COVID-19 Syndrome.

DETAILED DESCRIPTION:
Introduction: COVID-19 is an emerging pandemic disease caused by severe acute respiratory syndrome (SARS-CoV-2). Although most patients infected with SARS-CoV-2 are asymptomatic or have mild symptoms, some patients develop severe symptoms that can long-term impair their quality of life and functional capacity. SARS-CoV-2 is closely related to severe acute respiratory syndrome (SARS) with direct and indirect effects on several systems, especially the musculoskeletal system, in addition to the respiratory system. Some of these symptoms persist for a long time, called Post-COVID-19 Syndrome, directly interfering with the functional capacity and quality of life of these patients. Pilates exercises focus on breathing, postural symmetry, trunk stabilization, flexibility, joint mobility and strengthening through the full range of motion of all joints and not isolated muscle groups. Objectives: The objective of this study will be to evaluate the clinical and functional effects of a Pilates exercise program for patients with Post-Covid-19 syndrome after a period of intensive care admission and invasive mechanical ventilation. Methods: The study will be a clinical, randomized and controlled trial. 48 patients of both sexes, over 18 years of age, who have developed the severe form of COVID-19 and required at least 7 days of invasive mechanical ventilation will be recruited. Patients who currently require supplemental oxygen at home and who present motor, cognitive or neurological alterations that prevent the practice of Pilates will be excluded. They will be previously randomized in a 1:1 ratio by electronic system and blindly allocated to the intervention group that will perform an exercise protocol based on the Pilates method, 2x/week, for 12 weeks in therapeutic sessions of identical protocols lasting 60 min. All patients will be evaluated before and after for six minutes walk distance test, peripheral and respiratory muscle strength and endurance, post-COVID-19 functional status, dyspnea, fatigue and quality of life. The analysis of the data obtained during the research was carried out by an independent statistician who had access to the coded data and were based on intention-to-treat principles. Missing data will be assumed to be completely missing by chance. Multiple imputation was used to explain these missing data (STERNE et al., 2009). Missing values in the outcome variables were estimated using multiple imputation by chained equations after 50 imputed replicated data sets. Variables included in the multiple imputation process included (1) group factor, (2) time factor, and (3) the respective outcome variable. Descriptive statistics will be used to present the characteristics of participants in the two treatment groups. P values less than 0.05 will be considered to indicate statistical evidence of significance. The variables of fatigue, peripheral muscle strength, functional capacity, post-COVID functional status and HRQoL were analyzed using linear models of repeated measures (participants and time as random factors) which included all values measured after randomization with baseline scores and treatment clusters as covariates. Adjusted mean differences will be tested 12 weeks after randomization and start of intervention. Multiple comparisons were performed using the Tukey Test with p-values adjusted using the Holm procedure. Baseline variables were evaluated as predictors and moderators of treatment effects, including terms and interaction models. Effect sizes for primary and secondary endpoints were calculated as Cohen's d from estimated marginal means (SMD) and standard error estimates from the adjusted primary analysis. Effect sizes were interpreted according to Cohen's criteria (small ≤0.2; moderate=0.5; large ≥0.8)(COHEN, 1988). All analyzes were performed using RStudio version 0.99.486. Results: The expected results are based on the alternative hypothesis that Pilates exercises are clinically effective, improving functional performance, exercise tolerance, reducing symptoms and improving the quality of life of patients with symptoms of Post-COVID-19 Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously diagnosed with COVID-19, who required hospitalization and required invasive mechanical ventilation for at least 7 days and who were discharged between August and December 2021 to minimize regression to mean;
2. Both sexes;
3. Over 18 years of age.

Exclusion Criteria:

1. Need for supplemental home oxygen;
2. Motor or neurological or cognitive alteration that contraindicates the practice of Pilates.
3. Persistence of clinical signs of deep vein thrombosis
4. Upper limb dynamometry < 14 kgs for men and < 7 kgs for women would indicate very marked peripheral muscle weakness and would therefore contraindicate Pliates at the moment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | 12 weeks
  Functional capacity will be measured by the distance covered in the 6-minute walk test. The distance covered will be expressed in meters and compared in absolute and relative values to predict normality for the studied population.
Functional Status | 12 weeks
  Functional status will be measured by the Post-COVID-19 Functional Status scale,which is graded from 0 to 4, with the highest score being the worst.

SECONDARY OUTCOMES:
Peripheral muscle endurance | 12 weeks
  The peripheral muscle endurance test will be performed using the constant load test, with the time to exhaustion as the variable of interest.
Respiratory muscle strength | 12 weeks
  Respiratory muscle strength will be measured by isometric measurement of maximal respiratory pressures. The maximum respiratory pressures will be measured by a digital manovacuometer, and the measurement used for analysis will be expressed in cmH2O and considered as the highest value sustained for 1s
Peripheral muscle strength | 12 weeks
  Peripheral muscle strength will be measured by the manual grip test on the dominant upper limb and by the 1-repetition maximum test (1-RM) for the quadriceps on the same side. The measure used will be expressed in kilograms, as the largest load carried out.
Dyspnea | 12 weeks
  Dyspnea will be measured using the modified medical research council scale, graded from 0 to 4, with the highest value being the worst
Health-related quality of life | 12 weeks
  Health-related quality of life will be measured by the global score of the short form - 36. This questionnaire is scored from 0 to 100, with the higher the value, the better the health-related quality of life.questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle de Aguiar Zacaria, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro de Fisiatria e Reabilitação da Polícia Militar do Estado do Rio de Janeiro, Rio de Janeiro, Brazil

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT05722730/Prot_SAP_ICF_000.pdf